CLINICAL TRIAL: NCT05814809
Title: Phase I Study to Evaluate the Safety and Pharmacokinetics of JP-1366 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Evaluate the Safety and Pharmacokinetics of JP-1366 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-104
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): R → Washout period(7days) → T
  Interventions: Drug: JP-1366 20mg tablet; Drug: JP-1366 20mg capsule
- Sequence B (Experimental): T → Washout period(7days) → R
  Interventions: Drug: JP-1366 20mg tablet; Drug: JP-1366 20mg capsule

INTERVENTIONS:
Drug: JP-1366 20mg tablet — T : JP-1366 20mg tablet
  Other Names: Zastaprazan 20mg
Drug: JP-1366 20mg capsule — R : JP-1366 20mg capsule
  Other Names: Zastaprazan 20mg

SUMMARY:
To evaluate the safety and the pharmacokinetics of the JP-1366 20 mg tablet and capsule oral administration in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 19 years of age
2. Subjects who weigh ≥ 50 kg (or ≥ 45 kg in the case of females) with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2

Exclusion Criteria:

1. Subjects with clinically significant diseases or a medical history related to the digestive system, cardiovascular system, endocrine system, respiratory system, blood and tumor, infections diseases, kidney and urinary system, psychiatric and nervous system, musculoskeletal system, immune system, otorhinolaryngology, skin, and ophthalmological system
2. Subjects who have a history of gastrointestinal surgery (except simple appendectomy or herniotomy) or have gastrointestinal disorders that may affect the absorption of the drug
3. Subjects who received inducers or inhibitors of drug metabolizing enzymes
4. Subjects who have hypersensitivity to this drug, ingredients of this drug, or benzimidazoles, or have a medical history thereof
5. Patients receiving drugs containing atazanavir, nelfinavir, or rilpivirine
6. Subjects who are judged ineligible to participate in this study by the principal investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
AUCt of Zastaprazan(JP-1366 20mg) | Pre-dose(0 hour) and up to 34 hours in each period
Cmax of Zastaprazan(JP-1366 20mg) | Pre-dose(0 hour) and up to 34 hours in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Yangji Hospital, Seoul, South Korea